CLINICAL TRIAL: NCT01020409
Title: INFLACOR (INFLA-mmation A-fter C-ardiac O-pe-R-ation) - Use of Selected Genetic Variants, Cytokines, and Physiologic Parameters in the Prognosis of Postoperative Complications in Patients Undergoing Cardiopulmonary Bypass Cardiac Surgery
Brief Title: INFLACOR - Clinical and Genetic Predictors of Inflammation Related Complications After Heart Surgery
Acronym: INFLACOR
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Principal Investigator, Maciej M. Kowalik, Dr., Medical University of Gdansk
Other Study IDs: N N403 1815 34; MUG grant G-35 (Other: Medical University of Gdańsk)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: cardiac surgery; cardiopulmonary bypass; acute lung injury; acute respiratory distress syndrome; acute kidney injury; atrial fibrillation; postoperative psychosis; myocardial infarct; sepsis
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Acute Lung Injury; Respiratory Distress Syndrome; Acute Kidney Injury; Atrial Fibrillation; Myocardial Infarction; Sepsis | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, and blood morphologic elements after centrifugation frozen to -75C.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cardiac surgery with CPB use: Adult patients, who signed the informed consent, intervention: first-time scheduled heart surgery with CPB use.
  Interventions: Procedure: cardiac surgery with CPB use

INTERVENTIONS:
Procedure: cardiac surgery with CPB use — cardiac surgery with CPB use or ascending aorta surgery performed with use of cardiopulmonary bypass with or without aortic cross clamping.
  Other Names: heart valve surgery; open heart surgery

SUMMARY:
The aim of the study is to evaluate a clinically and economically most effective diagnostic algorithm for prediction of inflammatory response related complications in patients undergoing heart surgery with use of cardiopulmonary bypass.

DETAILED DESCRIPTION:
Identified so far predictors of mortality and/or morbidity in patients who undergo heart surgery with cardiopulmonary bypass (CPB), used in previous risk prediction models (EUROSCORE, CABDEAL, Cleveland), will be compared with new candidate variables:

1. anamnestic: recent tooth extractions, chronic inflammatory diseases, specific drug use;
2. biochemical: C-reacting protein, interleukin-6, tumor necrosing factor alpha;
3. genetical: single nucleotide polymorphisms of 10 genes associated with inflammatory response; and
4. clinical from the 1. postoperative day: systemic inflammatory response syndrome, APACHE-III score;

against their predictive capability of selected clinical phenotypes of inflammatory response occuring after surgery, beginning from day 2. after surgery.

ELIGIBILITY:
Inclusion Criteria:

* adults (age >=18)
* given and signed informed consent
* no previous cardiac surgery with opening the pericardium

Exclusion Criteria:

* previous cardiac surgery with opening the pericardium
* consent refused or not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (at least age 18), who signed informed consent, scheduled for elective cardiac surgery with use of cardiopulmonary bypass.
Sampling Method: Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Clinical phenotypes of inflammatory response: SIRS, acute lung injury/acute respiratory distress syndrome, acute kidney injury, atrial fibrillation, postoperative psychosis, perioperative myocardial infarct/injury, sepsis. | between day 2 after operation and hospital discharge

SECONDARY OUTCOMES:
all cause inhospital mortality | from day 2 after operation

CONTACTS AND LOCATIONS:
Overall Officials: Romuald Lango, MD, PhD, Study Chair — Medical University of Gdansk; Maciej M Kowalik, MD, PhD, Study Director — Medical University of Gdansk; Jan Rogowski, MD, PhD, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdańsk, Academic Clinical Centre, Department of Cardiac Anaesthesiology, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes
IPD can be made available to other researcher upon reasonable request.

REFERENCES:
- [Background] Butler J, Baigrie RJ, Parker D, Chong JL, Shale DJ, Pillai R, Westaby S, Rocker GM. Systemic inflammatory responses to cardiopulmonary bypass: a pilot study of the effects of pentoxifylline. Respir Med. 1993 May;87(4):285-8. doi: 10.1016/0954-6111(93)90024-t. PMID 9728228
- [Background] Asimakopoulos G. Mechanisms of the systemic inflammatory response. Perfusion. 1999 Jul;14(4):269-77. doi: 10.1177/026765919901400406. PMID 10456781
- [Background] Higgins TL, Estafanous FG, Loop FD, Beck GJ, Blum JM, Paranandi L. Stratification of morbidity and mortality outcome by preoperative risk factors in coronary artery bypass patients. A clinical severity score. JAMA. 1992 May 6;267(17):2344-8. PMID 1564774
- [Background] Nashef SA, Roques F, Michel P, Gauducheau E, Lemeshow S, Salamon R. European system for cardiac operative risk evaluation (EuroSCORE). Eur J Cardiothorac Surg. 1999 Jul;16(1):9-13. doi: 10.1016/s1010-7940(99)00134-7. PMID 10456395
- [Background] Kurki TS, Jarvinen O, Kataja MJ, Laurikka J, Tarkka M. Performance of three preoperative risk indices; CABDEAL, EuroSCORE and Cleveland models in a prospective coronary bypass database. Eur J Cardiothorac Surg. 2002 Mar;21(3):406-10. doi: 10.1016/s1010-7940(02)00007-6. PMID 11888755
- [Background] Butler J, Chong GL, Baigrie RJ, Pillai R, Westaby S, Rocker GM. Cytokine responses to cardiopulmonary bypass with membrane and bubble oxygenation. Ann Thorac Surg. 1992 May;53(5):833-8. doi: 10.1016/0003-4975(92)91446-g. PMID 1570980
- [Background] Lamm G, Auer J, Weber T, Berent R, Ng C, Eber B. Postoperative white blood cell count predicts atrial fibrillation after cardiac surgery. J Cardiothorac Vasc Anesth. 2006 Feb;20(1):51-6. doi: 10.1053/j.jvca.2005.03.026. PMID 16458214
- [Background] Podgoreanu MV, White WD, Morris RW, Mathew JP, Stafford-Smith M, Welsby IJ, Grocott HP, Milano CA, Newman MF, Schwinn DA; Perioperative Genetics and Safety Outcomes Study (PEGASUS) Investigative Team. Inflammatory gene polymorphisms and risk of postoperative myocardial infarction after cardiac surgery. Circulation. 2006 Jul 4;114(1 Suppl):I275-81. doi: 10.1161/CIRCULATIONAHA.105.001032. PMID 16820586
- [Background] Gaudino M, Di Castelnuovo A, Zamparelli R, Andreotti F, Burzotta F, Iacoviello L, Glieca F, Alessandrini F, Nasso G, Donati MB, Maseri A, Schiavello R, Possati G. Genetic control of postoperative systemic inflammatory reaction and pulmonary and renal complications after coronary artery surgery. J Thorac Cardiovasc Surg. 2003 Oct;126(4):1107-12. doi: 10.1016/s0022-5223(03)00396-9. PMID 14566255
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500
- [Background] Mitchell JD, Grocott HP, Phillips-Bute B, Mathew JP, Newman MF, Bar-Yosef S. Cytokine secretion after cardiac surgery and its relationship to postoperative fever. Cytokine. 2007 Apr;38(1):37-42. doi: 10.1016/j.cyto.2007.04.009. Epub 2007 Jun 14. PMID 17572096
- [Background] Bellomo R, Kellum JA, Ronco C. Defining and classifying acute renal failure: from advocacy to consensus and validation of the RIFLE criteria. Intensive Care Med. 2007 Mar;33(3):409-13. doi: 10.1007/s00134-006-0478-x. Epub 2006 Dec 13. PMID 17165018
- [Background] Bernard GR, Artigas A, Brigham KL, Carlet J, Falke K, Hudson L, Lamy M, Legall JR, Morris A, Spragg R. The American-European Consensus Conference on ARDS. Definitions, mechanisms, relevant outcomes, and clinical trial coordination. Am J Respir Crit Care Med. 1994 Mar;149(3 Pt 1):818-24. doi: 10.1164/ajrccm.149.3.7509706.
- [Background] Knaus WA, Wagner DP, Draper EA, Zimmerman JE, Bergner M, Bastos PG, Sirio CA, Murphy DJ, Lotring T, Damiano A, et al. The APACHE III prognostic system. Risk prediction of hospital mortality for critically ill hospitalized adults. Chest. 1991 Dec;100(6):1619-36. doi: 10.1378/chest.100.6.1619. PMID 1959406
- [Background] Gemert van LA, Schuurmans MJ. The Neecham Confusion Scale and the Delirium Observation Screening Scale: capacity to discriminate and ease of use in clinical practice. BMC Nurs. 2007 Mar 29;6:3. doi: 10.1186/1472-6955-6-3. PMID 17394635
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction. Universal definition of myocardial infarction. Eur Heart J. 2007 Oct;28(20):2525-38. doi: 10.1093/eurheartj/ehm355. No abstract available. PMID 17951287